CLINICAL TRIAL: NCT00019032
Title: PHASE I STUDY OF T-CELL LARGE GRANULAR LYMPHOCYTIC LEUKEMIA USING THE MIK-BETA 1 MONOCLONAL ANTIBODY DIRECTED TOWARD THE IL-2R BETA SUBUNIT
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064038; NCI-95-C-0054K; NCT00001425 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2004-04

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Large Granular Lymphocytic | interventions — Hu-Mik-beta-1 monoclonal antibody

INTERVENTIONS:
Biological: monoclonal antibody Mik-beta-1

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the toxicity of murine monoclonal antibody Mik-beta-1 (MOAB Mik-beta-1) in patients with T-cell large granular lymphocytic leukemia associated with granulocytopenia, anemia, or thrombocytopenia.
* Determine the clinical response in patients treated with this drug.
* Assess the effect of this drug on the number of circulating CD3+, CD8+ expressing granular lymphocytes and the number of polymorphonuclear leukocytes, red blood cells, and platelets in this patient population.
* Monitor patients for the time course of decline in circulating infused MOAB Mik-beta-1 and for the production of human antibodies to IV infused murine MOAB Mik-beta-1.

OUTLINE: This is a dose-escalation study.

Patients receive monoclonal antibody Mik-beta-1 (MOAB Mik-beta-1) IV over 2 hours on days 1, 4, 7, and 10. Patients achieving a complete response (CR) or partial response (PR) may receive 1 additional course beginning no sooner than 4 weeks after completion of the first course, in the absence of antibodies to MOAB Mik-beta-1. Treatment continues in the absence of disease progression, unacceptable toxicity, or severe allergic reaction.

Cohorts of 3-6 patients receive escalating doses of MOAB Mik-beta-1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 6-10 days and at 4-6 weeks after therapy. Patients with a PR or CR may be followed every 6 months for 2 years or until relapse. All patients are followed for survival.

PROJECTED ACCRUAL: A maximum of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed T-cell large granular lymphocytic (T-LGL) leukemia associated with clinically significant hematocytopenia demonstrated by one of the following values while off growth factor support:

  * Absolute neutrophil count less than 1,000/mm^3
  * Hemoglobin less than 8 g/dL
  * Platelet count less than 50,000/mm^3
* Clinically evaluable disease with peripheral blood T-LGL leukemia cells expressing the CD3+, CD8+ phenotype detectable by FACS
* Monoclonal T-cell population in peripheral blood (circulating mononuclear cells) demonstrated by TCR beta or gamma chain gene rearrangement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50-100%

Life expectancy:

* More than 2 months

Hematopoietic:

* See Disease Characteristics
* No active major bleeding episode within the past 4 weeks

Hepatic:

* Direct bilirubin less than 1.5 mg/dL

Renal:

* Creatinine less than 2.0 mg/dL

Other:

* No concurrent serious active infection
* Patients with fever without apparent site of infection may begin study while on antibiotics as long as the following are true:

  * No pathogenic organism in culture
  * Afebrile (maximum temperature less than 38°C) for at least 5 days
* HIV negative
* No other primary cancer other than basal cell skin cancer
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior interferon
* Concurrent filgrastim (G-CSF), sargramostim (GM-CSF), interleukin-11, or similar sustained-release/long-acting product (e.g., pegylated G-CSF) allowed if dose established at least 4 weeks prior to study participation
* No concurrent interferon

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* Concurrent corticosteroids allowed if dose established at least 3 weeks prior to study participation

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 1 week since completion of prior antibiotic regimen for serious infectious episode
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1996-03

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A. Waldmann, MD, Study Chair — NCI - Metabolism Branch;MET
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States